CLINICAL TRIAL: NCT01908595
Title: An Open-label, Multi-center, Long-term Study to Evaluate the Safety and Efficacy of M518101 in Subjects With Plaque Psoriasis
Brief Title: Long Term Study to Evaluate Safety and Efficacy of M518101 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M518101-US04
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- M518101 (Experimental): Proper quantity twice daily
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: M518101

SUMMARY:
This study is to evaluate the efficacy and safety for long term use of M518101 in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Who are able and willing to give signed informed consent
* Who are male or females aged 18 years or older with plaque psoriasis confirmed by the Investigator.
* Who have up to 20% of body surface area (BSA) afflicted with plaques
* Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

* Who have a history of allergy to vitamin D3 derivative preparations or a history of relevant drug hypersensitivity.
* Who are pregnant or lactating.
* Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
* Who are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
* Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study.
* Whose serum calcium levels exceed the upper limit of reference range
* Who have used any investigational medicinal product and/or participated in any clinical study within 60 days of treatment.
* Who have been treated with systemic therapy within 30days of treatment.
* Who have treated with biologics within 5 half-lives of the biologics before the day of treatment
* Who have been treated with topical therapy within 14days before the day of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time course change of Investigator Global Assessment | 4 weeks interval

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Agave Clinical Research, Mesa, Arizona
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Dermatology Research Associates, Los Angeles, California
  - Medical Center for Clinical Research, San Diego, California
  - ATS Clinical Research, Santa Monica, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Dermatology and Aesthetic Center Skin Care, Boca Raton, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - FXM Research Miramar, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Peachtree Dermatology Associates Research Center, Atlanta, Georgia
  - Northshore University Health System, Skokie, Illinois
  - South bend clinic, South Bend, Indiana
  - Kansas City Dermatology, Overland Park, Kansas
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - J Woodson Dermatology and Associates, Henderson, Nevada
  - New York University, New York, New York
  - PMG research of raleigh, Cary, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Bager Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - PMG Research of Bristol, Kingsport, Tennessee
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - The skin wellness center, Knoxville, Tennessee
  - Suzanne Bruce & Associates, Houston, Texas
  - Research Across America, Plano, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Stephen Miller, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Madison Skin & Research, Madison, Wisconsin